CLINICAL TRIAL: NCT04442373
Title: Impact of Surgical Injury on Global Haemostatic Tests in Patients Undergoing Total Hip Replacement With Subgroup Analysis of Patients With Bone Neoplasm. A Single-centre Observational Prospective Trial
Brief Title: Impact of Surgical Injury on Haemostatic Tests in Patients Undergoing Total Hip Replacement With Subgroup Analysis of Patients With Neoplasm
Acronym: I-SIGHT-THR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Jan Pluta, Principal Investigator, Medical University of Warsaw
Other Study IDs: ROTEM-THR
Record Dates: First submitted 2020-03-08; First posted 2020-06-22 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Total Hip Replacement; Thromboelastometry; Bone Neoplasm of Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing THR with no known bone neoplasm: Pre- and postoperative blood sampling for ROTEM assessment in THR patients
  Interventions: Diagnostic Test: Rotational thromboelastometry
- Patients undergoing THR with known bone neoplasm: Pre- and postoperative blood sampling for ROTEM assessment before and after THR in patients with bone neoplasm
  Interventions: Diagnostic Test: Rotational thromboelastometry

INTERVENTIONS:
Diagnostic Test: Rotational thromboelastometry — 1.8 ml blood sample
  Other Names: ROTEM

SUMMARY:
Total hip replacement (THR) is associated with extensive tissue injury and considerable blood loss that can be complicated by hyperfibrinolysis with an increased need for blood transfusion. THR in patients with cancer involving the hip joint, can reduce pain and improve or maintain the function and quality of life. However, these patients have an increased likelihood of haemostatic abnormalities, such as thrombosis or extensive blood loss. Rotational thromboelastometry is a point-of-care viscoelastic assay that can provide a measure of coagulation disorders in the above settings, and this is still under review. The objective of this prospective cohort study is to quantitate the changes in clot formation dynamics following THR with a subgroup analysis of patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing primary elective total hip replacement

Exclusion Criteria:

* Patients unable to consent to trial
* Active deep and superficial vein thrombosis
* Coagulopathy in initial coagulation screen tests
* Platelet count below 100 thousand
* Patients on antithrombotic medications (except prophylactic low molecular weight heparins and acetylsalicylic acid up to 75 mg per day)
* Preoperative haemoglobin < 10 g/dl
* Female patients who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective total hip replacement
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
INTEM parameters change from preoperative to postoperative values | 30 minutes before and 30 minutes after surgery
EXTEM parameters change from preoperative to postoperative values | 30 minutes before and 30 minutes after surgery
FIBTEM parameter change from preoperative to postoperative values | 30 minutes before and 30 minutes after surgery

SECONDARY OUTCOMES:
Total volume of infused fluids | From first fluid on day of surgery to end of surgery, an average of 12 hours
  Crystalloids, blood products
Pre- and postoperative haemoglobin and haematocrit | From day before surgery to postoperative day 3
Intraoperative blood loss | Blood loss as measured during surgery
  Amount of blood loss in millilitres
Hip Disability and Osteoarthritis Outcome Score (HOOS) | The day before surgery and at 6 ± 1 months, 12 ± 1 month after surgery
  Instrument for measuring outcome following surgery with higher scores representing better function. Score from 0 to 100.
The 36-Item Short Form Health Survey (SF-36) | The day before surgery and at 6 ± 1 months, 12 ± 1 month after surgery
  Health related Quality of Life measure. Higher score indicates better health state with eight scaled scores each from 0 to 100.
Visual Analogue Scale (VAS) score | The day before surgery and at 6 ± 1 months, 12 ± 1 month after surgery
  The ends of the scale are defined as the extreme limits of the pain. Orientated from the left (no pain) to the right (worst imaginable pain) measured in millimeters from 0 to 100.

OTHER OUTCOMES:
Rate of thrombotic events | up to 12 months after surgery
  Pulmonary embolism, deep and superficial vein thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Jan Pluta, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- I Department of Anesthesiology and Intensive Care Warsaw Medical University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided